CLINICAL TRIAL: NCT00004468
Title: Study of Topical Calcitriol or Oral Calcitriol in Patients With Psoriasis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funds
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Boston University (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 199/13927; BUSM-87-011 (Other: Boston University School of Medicine); R01DK043690 (NIH)
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Psoriasis
Keywords: dermatologic disorders; psoriasis; rare disease
MeSH Terms: conditions — Psoriasis; Skin Diseases; Rare Diseases | interventions — Calcitriol

INTERVENTIONS:
Drug: calcitriol

SUMMARY:
OBJECTIVES: I. Evaluate the long term safety and efficacy of orally administered calcitriol in patients with at least 5% of their body covered with psoriasis.

II. Evaluate the long term safety and efficacy of topically administered calcitriol in patients with at least 5% of their body covered with psoriasis.

III. Compare the topical calcitriol treatment to the oral calcitriol treatment in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a part placebo-controlled (arm I) study. Patients either apply topical petrolatum (Vaseline) with calcitriol (vitamin D3) on a psoriatic lesion daily and petrolatum only on an other similar lesion daily to serve as a control (arm I) or receive oral calcitriol nightly (arm II).

Arm I patients continue treatment for at least 2 months. At the end of 2 months of topical treatment, one biopsy is taken of the lesion treated with calcitriol, one biopsy of the lesion treated with petrolatum alone, and one biopsy of skin unaffected by psoriasis. Lesions are also photographed prior to therapy, 2-4 weeks during therapy for the first two months, then once every 1-3 months, and then once at end of treatment.

Arm II patients increase dosage of oral calcitriol every 2 weeks up to a maximum dosage daily in the absence of adverse effects (high urinary calcium or serum calcium levels). Patients continue treatment for at least 1 month. Lesions are photographed prior to therapy, 2-4 weeks during therapy, and then once at end of treatment.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Psoriasis covering at least 5% of body

--Prior/Concurrent Therapy--

At least 30 days since prior systemic therapy for psoriasis

At least 14 days since prior topical therapy for psoriasis

No other concurrent treatment for psoriasis for the first 2-4 months of study

No calcium supplement greater than 1,000 mg per day

--Patient Characteristics--

No hypercalcemia

No hypercalciuria

Not pregnant

Effective contraception required of all fertile patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1998-10

CONTACTS AND LOCATIONS:
Overall Officials: Michael F. Holick, Study Chair — Boston University